CLINICAL TRIAL: NCT06143059
Title: Sex and Sex Hormone Factors Influencing Acute Alcohol Effects on Sleep Physiology
Brief Title: The Effects of Sex Hormones and Alcohol on Sleep
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: PI transferring work elsewhere
Sponsor: Lauren Whitehurst (Other)
Collaborators: Ohio State University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Lauren Whitehurst, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 77098; R01AA030308 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
Keywords: Sex hormones; Sleep disruption
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Women will complete one alcohol-placebo session pair during the mid-follicular phase of the menstrual cycle and one pair during the late luteal phase. Men will complete two session pairs at matched intervals.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the nurse administering the IV alcohol or saline will know which one has been administered
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Alcohol Administration - Late Luteal Phase (Experimental): During the late luteal phase of a female participant's menstrual cycle, participants will complete a lab session where alcohol is administered intravenously. The infusion will include a 30-minute linear ascension from 0mg% breath alcohol content (BrAC) to 100mg%, followed by a 60-minute 'clamping' of BrAC at 100mg%. Subjects will then be monitored while they sleep, using polysomnography. Male subjects will complete this and the placebo session at intervals that are matched to the female subjects. The placebo and alcohol sessions during late luteal phase will take place 1-2 days apart, and their order will be randomized.
  Interventions: Drug: Ethanol
- Placebo - Late Luteal Phase (Placebo Comparator): During the late luteal phase of a female participant's menstrual cycle, participants will complete a lab session where saline is administered intravenously, as placebo, for 90 minutes. Subjects will then be monitored while they sleep, using polysomnography. Male subjects will complete this and the experimental session at intervals that are matched to the female subjects. The placebo and alcohol sessions during late luteal phase will take place 1-2 days apart, and their order will be randomized.
  Interventions: Drug: Saline
- Alcohol Administration - Mid-Follicular Phase (Experimental): During the mid-follicular phase of a female participant's menstrual cycle, participants will complete a lab session where alcohol is administered intravenously. The infusion will include a 30-minute linear ascension from 0mg% breath alcohol content (BrAC) to 100mg%, followed by a 60-minute 'clamping' of BrAC at 100mg%. Subjects will then be monitored while they sleep, using polysomnography. Male subjects will complete this and the placebo session at intervals that are matched to the female subjects. The placebo and alcohol sessions during mid-follicular luteal phase will take place 1-2 days apart, and their order will be randomized.
  Interventions: Drug: Ethanol
- Placebo - Mid-Follicular Phase (Placebo Comparator): During the mid-follicular phase of a female participant's menstrual cycle, participants will complete a lab session where saline is administered intravenously, as placebo, for 90 minutes. Subjects will then be monitored while they sleep, using polysomnography. Male subjects will complete this and the experimental session at intervals that are matched to the female subjects. The placebo and alcohol sessions during mid-follicular phase will take place 1-2 days apart, and their order will be randomized.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ethanol — Sterile, 95% ethanol will be administered through IV infusion
  Arms: Alcohol Administration - Late Luteal Phase; Alcohol Administration - Mid-Follicular Phase
Drug: Saline — Saline is administered as the placebo
  Arms: Placebo - Late Luteal Phase; Placebo - Mid-Follicular Phase

SUMMARY:
Rates of heavy drinking and Alcohol Use Disorder (AUD) are increasing in women, but research on alcohol-related harms in women - including alcohol's impact on sleep - has been minimal. Numerous studies in men show that alcohol impairs sleep, and preliminary evidence suggests that women may be even more sensitive to alcohol-disrupted sleep due to their sex hormones, which fluctuate across both their menstrual cycles and their reproductive lifespans.

This study will investigate the influence of sex, menstrual cycle phase, and sex hormones on alcohol-disrupted sleep in adults ages 21-45. Healthy women and men will complete two sets of placebo-controlled lab sessions, during the mid-follicular and late luteal phases of female participants' menstrual cycles. During these sessions, participants will receive a dose of alcohol or a placebo (saline) and they will then be monitored (with polysomnography) while they sleep. At-home sleep and alcohol use will also be measured through actigraphy, daily sleep and wake diaries, and alcohol wrist sensors.

Investigators hypothesize that women will show greater disruption of sleep following alcohol use or administration than men, and that alcohol-disrupted sleep will be more pronounced in the late luteal phase compared to the mid-follicular phase. Investigators also expect that estradiol will be negatively associated with alcohol-disrupted sleep, whereas progesterone will be positively associated with alcohol-disrupted sleep.

DETAILED DESCRIPTION:
Rates of heavy drinking and Alcohol Use Disorder (AUD) are increasing in women at an alarming pace. Such drastic increases in drinking will have a significant negative impact on women's health. Unfortunately, until recently heavy drinking has been considered a male-oriented problem, and consequently research on alcohol-related harms in women has been minimal. One specific aspect of women's health that may be negatively affected by alcohol is sleep. Numerous studies in men show that although alcohol has an initial sedative effect, it leads to frequent awakenings and impaired rapid eye movement sleep in the second half of the night.

Preliminary evidence suggests that women experience similar impairment, and that they may be even more sensitive to alcohol-disrupted sleep than men. Further, in the general population, women are at greater risk for insomnia and sleep disturbances than men, in part because women's sleep is sensitive to fluctuations in ovarian hormones. Hormonal influences on sleep are especially pronounced in older women of late reproductive age. However, the influence of sex and sex hormones on alcohol-disrupted sleep across the reproductive lifespan in women is unknown.

Here, investigators will determine the influence of sex, menstrual cycle phase, and sex hormones on alcohol-disrupted sleep in adults across the reproductive age range for women. Healthy women and men (age 21-45) will complete two pairs of experimental sessions in which they receive a dose of alcohol (target breath alcohol content [BrAC] = 100mg%, intravenous) or placebo (saline) one hour prior to eight hours of polysomnographically-monitored sleep in the lab. Women will complete one alcohol-placebo session pair during the mid-follicular phase of the menstrual cycle and one pair during the late luteal phase. Men will complete two session pairs at matched intervals. Participants will also complete two 5-day at-home monitoring periods of naturalistic sleep and alcohol consumption patterns during the mid-follicular and late luteal phases. Sleep and alcohol use will be assessed with actigraphy, daily sleep and wake diaries, and alcohol wrist sensors.

Investigators hypothesize that women will show greater disruption of sleep following alcohol than men and that alcohol-disrupted sleep, measured in lab with polysomnography and at-home with actigraphy, will be more pronounced in the late luteal phase compared to the mid-follicular phase. Investigators also expect that estradiol will be negatively associated with alcohol-disrupted sleep, whereas progesterone will be positively associated with alcohol-disrupted sleep.

This study will provide essential information regarding alcohol effects on sleep across the reproductive age span in women, and critically, how these effects are moderated by sex, menstrual cycle, and fluctuations in sex hormones. Findings will directly inform future interventions aimed at reducing alcohol consumption and the negative impacts of alcohol on sleep in women. Given the wide-ranging impact of sleep on other areas of function, including cognition, stress, and well-being, such interventions will have a substantial positive impact on women's health.

ELIGIBILITY:
Inclusion Criteria:

* 21-45 years old
* At least a high school education
* Fluency in English
* Report drinking at least twice per week and at least weekly binge episodes (4/5+ drinks for women/men in a 2-hour period)
* Regular ovulatory menstrual cycles (21-35 days in length) for women

Exclusion Criteria:

* Any serious medical problems (e.g., liver disease, cardiac abnormality/arrhythmia, pancreatitis, diabetes, neurological problems, gastrointestinal disorders, hypertension, and congestive heart failure)
* Any clinical sleep disorder, including insomnia and obstructive sleep apnea (OSA)
* Any psychiatric condition that could affect sleep/wake cycles (including major depression, generalized anxiety disorder, bipolar disorder, and post-traumatic stress disorder)
* Any medication use that is likely to affect sleep/wake function or cardiovascular functioning (including antidepressants, anxiolytic or soporific medication, and beta-blockers)
* Taking medication for which alcohol consumption is contraindicated
* Substance use disorder other than mild or moderate alcohol use disorder
* Positive urine screen for illegal drugs other than cannabis
* Currently seeking or past-12-month history of inpatient or intensive treatment for addictive behaviors
* Pregnancy, nursing or planning to become pregnant in the next 3 months for women
* Use of hormonal contraception or planning to begin use of hormonal contraception in the next 3 months for women
* Reports smoking > 5 cigarettes per day (to avoid acute nicotine effects or withdrawal during experimental sessions)
* Has flushing response to alcohol
* Works the night shift

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Slow Wave Sleep Minutes | Night 1 (alcohol administration, late luteal phase; 8 hours)
  Number of minutes participants spend in slow wave sleep during the night
Slow Wave Sleep Minutes | Night 2 (placebo, late luteal phase; 8 hours)
  Number of minutes participants spend in slow wave sleep during the night
Slow Wave Sleep Minutes | Night 3 (alcohol administration, mid-follicular phase; 8 hours)
  Number of minutes participants spend in slow wave sleep during the night
Slow Wave Sleep Minutes | Night 4 (placebo, mid-follicular phase; 8 hours)
  Number of minutes participants spend in slow wave sleep during the night
Rapid Eye Movement Sleep Minutes | Night 1 (alcohol administration, late luteal phase; 8 hours)
  Number of minutes participants spend in rapid eye movement (REM) sleep during the night
Rapid Eye Movement Sleep Minutes | Night 2 (placebo, late luteal phase; 8 hours)
  Number of minutes participants spend in rapid eye movement (REM) sleep during the night
Rapid Eye Movement Sleep Minutes | Night 3 (alcohol administration, mid-follicular phase; 8 hours)
  Number of minutes participants spend in rapid eye movement (REM) sleep during the night
Rapid Eye Movement Sleep Minutes | Night 4 (placebo, mid-follicular phase; 8 hours)
  Number of minutes participants spend in rapid eye movement (REM) sleep during the night
Wake After Sleep Onset | Night 1 (alcohol administration, late luteal phase; 8 hours)
  Number of one minute arousal epochs after sleep was initiated during the night
Wake After Sleep Onset | Night 2 (placebo, late luteal phase; 8 hours)
  Number of one minute arousal epochs after sleep was initiated during the night
Wake After Sleep Onset | Night 3 (alcohol administration, mid-follicular phase; 8 hours)
  Number of one minute arousal epochs after sleep was initiated during the night
Wake After Sleep Onset | Night 4 (placebo, mid-follicular phase; 8 hours)
  Number of one minute arousal epochs after sleep was initiated during the night
Sleep Efficiency | Night 1 (alcohol administration, late luteal phase; 8 hours)
  Amount of time spent asleep / amount of time in bed *100
Sleep Efficiency | Night 2 (placebo, late luteal phase; 8 hours)
  Amount of time spent asleep / amount of time in bed *100
Sleep Efficiency | Night 3 (alcohol administration, mid-follicular phase; 8 hours)
  Amount of time spent asleep / amount of time in bed *100
Sleep Efficiency | Night 4 (placebo, mid-follicular phase; 8 hours)
  Amount of time spent asleep / amount of time in bed *100

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Whitehurst, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States